CLINICAL TRIAL: NCT03738267
Title: Study on the Occurrence of Head and Neck Cancers During Pregnancy
Acronym: REFCORbirth
Status: Suspended | Type: Observational
Why Stopped: number of inclusions not reached
Sponsor: Centre Francois Baclesse (Other)
Collaborators: French scientific group REFCOR (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-A01220-55
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Pregnancy Related
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Head and neck cancers that occurred during pregnancy

ELIGIBILITY:
Inclusion Criteria:

* 18 year old woman or over at the time of participation
* PS 0 -2
* Cancer diagnosed (biopsy date) from 01/01/2010 between the second week of pregnancy and the 12 months postpartum.
* Primitive may concern the following sites:

oral cavity, nasopharynx, oropharynx, hypopharynx, larynx, prevalent lymphadenopathy, nasal cavity, salivary glands, dental tumors, ear tumors, paragangliomas optic pathways, facial sinus / facial mass, nose, ear and other head and neck

* All histologies (epithelial tumors, sarcomas, mucosal melanomas, embryonic tumors, undifferentiated tumors)
* Patient receiving or having received a specific oncological treatment among surgery, radiotherapy, chemotherapy, hormone therapy.
* All stages allowed: localized stages and metastatic stages immediately.
* No opposition of the patient to participate in this study

Exclusion Criteria:

* Any other neoplastic antecedent
* Exclusion of metastases at the level of the VADS of another primitive than a cancer of the VADS
* Exclusion of hematological tumors (lymphoma) and glial tumors
* Person subject to a legal protection measure or unable to express their consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancers of Head and Neck that occurred during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Serological status of patients | Through study completion, an average of 5 years
  Number of patients with positive or negative serological status for PVH (Papilloma Virus Humain) and EBV (Epstein-Barr Virus)
Characteristics pregnancy of patients | Through study completion, an average of 5 years
  Presence or absence of maternal-fetal diseases
Tumor characteristics of patients | Through study completion, an average of 5 years
  Histological type of cancer
Tumor characteristics of patients | Through study completion, an average of 5 years
  Localization of cancer

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Chu Besancon, Besançon
  - Chu Bordeaux, Bordeaux
  - Centre François Baclesse, Caen
  - Chu Grenoble Alpes, Grenoble
  - Ap-Hp Tenon, Paris
  - Chu Poitiers, Poitiers
  - Chu Toulouse, Toulouse
  - Institut Gustave Roussy IGR, Villejuif